CLINICAL TRIAL: NCT04340726
Title: Periimplant Bone Changes in Different Abutment Heights and Insertion Timing in Posterior Mandibular Areas: Results From a Randomized Prospective Clinical Trial
Brief Title: Periimplant Bone Changes in Different Abutment Heights and Insertion Timing in Posterior Mandibular Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Católica Portuguesa (Other)
Responsible Party: Principal Investigator, Tiago Borges, Professor, Universidade Católica Portuguesa
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 02/2015
Record Dates: First submitted 2020-04-03; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: One time abutment

SUMMARY:
The aim of this study was to compare the influence of the abutment height and insertion timing on early marginal bone loss (MBL) in posterior mandibular partial implant-supported restorations.

Material and methods: The study was planned as a prospective, randomized, controlled parallel group including subjects in need of two implants for the restoration of an edentulous posterior mandibular area. Data were gathered on age, gender, attached gingiva height, bleeding on probing (BoP), smoking habits and previous periodontitis. The patients were allocated into three groups: Group A implants were immediately connected to 2 mm height abutments; Group B implants were immediately connected to 1 mm height abutments; Group C implants were left to heal in a sub-mucosal position and 2 mm abutments were inserted in a second stage surgery. Peri-apical radiographs were taken at the implant surgery (baseline), 4 weeks after surgery (T1), 16 weeks after implant placement at the final restoration delivery (T2) and 1-year after implant placement (T3).

ELIGIBILITY:
Inclusion Criteria:

* patients age > 18 years;
* American Society of Anaesthesiologists (ASA) status I;
* no systemic medication or condition known to potentially alter bone metabolism; - absense of acute periodontal condition.

Exclusion Criteria:

* lack of primary stability at implant surgery;
* need for bone regeneration procedures during surgery;
* inability to correct place the implant in accordance with the prosthetic requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Marginal bone changes | 60 months
  Crestal bone changes that occur around the dental implant

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Católica Portuguesa, Viseu, Portugal